CLINICAL TRIAL: NCT05163834
Title: A Randomized, Open-label, Placebo-Controlled, Parallel-Group Study to Evaluate the Immune Response to the Polyvalent Pneumococcal Vaccine (PNEUMOVAX 23) in Healthy Participants Receiving Intravenous Efgartigimod or Placebo
Brief Title: Immune Response to PNEUMOVAX 23 in Healthy Adults Receiving Efgartigimod IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ARGX-113-2102; 2021-004878-53 (EudraCT Number)
Record Dates: First submitted 2021-11-23; First posted 2021-12-20 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — efgartigimod alfa; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Efgartigimod-1 (Experimental): Weekly efgartigimod infusions and the pneumovax 23 vaccine on day 22
  Interventions: Biological: Efgartigimod; Biological: PNEUMOVAX 23
- Efgartigimod-2 (Experimental): Weekly efgartigimod infusions and the pneumovax 23 vaccine on day 36
  Interventions: Biological: Efgartigimod; Biological: PNEUMOVAX 23
- Placebo (Placebo Comparator): Weekly placebo infusions and the pneumovax 23 vaccine on day 22
  Interventions: Other: Placebo; Biological: PNEUMOVAX 23

INTERVENTIONS:
Biological: Efgartigimod — intravenous infusion of efgartigimod
  Arms: Efgartigimod-1; Efgartigimod-2
Other: Placebo — intravenous infusion of placebo
  Arms: Placebo
Biological: PNEUMOVAX 23 — PNEUMOVAX 23 vaccine

SUMMARY:
This is a randomized, open-label, placebo-controlled phase 1 study in healthy adult volunteers to provide information regarding vaccination with a common pneumococcal polysaccharide vaccine while receiving efgartigimod.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the informed consent form (ICF)
* Healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body mass index (BMI) between 18 kg/m2 to 30 kg/m2 (inclusive)
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants must agree not to donate sperm from the time the ICF was signed until the end of the study
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before study intervention can be administered.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
* Abstains from smoking for at least 3 months prior to screening
* Negative urine drug screen and negative alcohol urine test
* Agrees to restrict excessive strenuous physical activities 96 hours prior to screening, 96 hours prior to the visits in the treatment period, and 96 hours prior to the visits in follow-up period.

Exclusion Criteria:

* Clinically significant active or chronic bacterial, viral, including or fungal infection at day -1
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of study intervention. Participants with the following cancers can be included at any time: Adequately treated basal cell or squamous cell skin cancer ; Carcinoma in situ of the cervix and Carcinoma in situ of the breast; Incidental histological finding of prostate cancer (TNM stage T1a or T1b).
* Clinical evidence of other significant serious diseases, a recent major surgery, or any other condition that, in the opinion of the investigator, could confound the results of the study or put the participant at undue risk
* Use of an investigational product within 2 months or 5 half-lives (whichever is longer) before the first dose of study intervention; Use of any monoclonal antibody within 3 months prior to the initial study intervention administration; Use of any systemic immunosuppressant agent within 6 months prior to the initial study intervention administration; Use of any systemic steroid within 3 months prior to the initial study intervention administration; Use of B-cell depleting agents in the year before the initial screening visit
* Previously participated in a clinical study with efgartigimod and received at least 1 dose of efgartigimod
* Positive serum test screening for an active viral infection with any of the following conditions: Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human immunodeficiency virus (HIV) based on test results that are associated with an acquired immunodeficiency syndrome (AIDS)-defining condition, or a CD4 count ≤200 cells/mm3.
* Positive nasopharyngeal swab antigen test for SARS-CoV-2 on day -1. Any contact with SARS-CoV-2 positive or COVID-19 patients within the last 2 weeks prior to admission.
* Total IgG ≤6 g/L at screening
* Current or history of (ie, within 12 months of screening) alcohol, drug, or medication abuse
* Known hypersensitivity reaction to any of the excipients of study intervention, the PNEUMOVAX 23 vaccine, or any of its excipients
* Pregnant or lactating females and those who intend to become pregnant during the study or within 90 days after the last dose of study intervention
* Received a live or live-attenuated vaccine less than 4 weeks before screening. The receipt of any inactivated, subunit, polysaccharide, or conjugate vaccine at any time before screening is not considered exclusionary
* Received a pneumococcal vaccine within the past 10 years
* Documented pneumococcal infection within the past 5 years prior to first administration of the study intervention
* Has a clinically relevant abnormality detected on ECG recording regarding either rhythm or conduction. A first-degree heart block or sinus arrhythmia will not be considered a significant abnormality.
* Had significant blood loss (including blood donation ≥500 mL) within 12 weeks prior to the (first) study intervention administration
* Has any condition impairing phlebotomy
* Is an employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as a family member of an employee or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Variation in the immune response assessed by comparing pneumococcal capsular polysaccharide (PCP) titers pre- and postadministration of the PNEUMOVAX 23 vaccine between study arms | throughout the study (up to 12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator site 1, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided